CLINICAL TRIAL: NCT04870346
Title: Long Term Follow-up Observational Study After Clinical Trials of AMG531 (Romiplostim) in Patients With Untreated Aplastic Anemia
Status: Active, not recruiting | Type: Observational
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 531-005
Record Dates: First submitted 2021-04-22; First posted 2021-05-03 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Aplastic Anemia
Keywords: aplastic anemia
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the long-term efficacy and safety after the end of romiplostim treatment by observation [up to 5 years] of patients who were registered for Study 531-003/531-004 in immunosuppressive therapy-naïve patients with aplastic anemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose written consent to participate in this research was obtained among patients registered for Study 531-003/531-004
* Of the patients who died before their consent to participate in this research was obtained among those registered for Study 531-003/531-004, patients whose legally authorized representatives such as their family had given the consent or patients whose legally authorized representatives had not refused in the disclosure of information by opt-out
* Of the patients who died before their consent to participate in this research was obtained among those registered for Study 531-003/531-004, patients, patients for whom the consent process exemption was approved by the Ethics Review Committee, etc. of the participating medical institutions at the participating medical institutions in the countries without the opt-out system

Exclusion Criteria:

* Patients who are judged by the investigator or sub-investigator to be unfavorable for participation in this research

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled in Study 531-003/531-004
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Hematological response at 2 years after the start of romiplostim treatment in Study 531-003/531-004 | 2 years
Hematological response at up to 5 years after the start of romiplostim treatment in Study 531-003/531-004 | 5 years

SECONDARY OUTCOMES:
The duration of hematological response, and the presence or absence of occurrence of new chromosomal abnormality or transformation to AML/MDS. | 52, 78, 104, 130, 156, 182, 208, 234, 260 weeks
  1. Duration of hematological response in patients who achieved hematologic response at the completion of Study 531-003/531-004
  2. Time courses of Hb level (g/dL)
  3. Time courses of platelet count (/μL)
  4. Time courses of neutrophil count (/μL)
  5. Presence or absence of platelet blood cell transfusion
  6. Presence or absence of red blood cell transfusion
  7. Presence or absence of G-CSF product administration
  8. Dose level and administration period of cyclosporine A
  9. Presence or absence of transformation to MDS/AML
  10. Presence or absence of occurrence of new chromosome abnormality
  11. Time to the start of subsequent treatment or to death
  12. Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Hirohito Yamazaki, Principal Investigator — Kanazawa University Hospital, Blood Transfusion Department
Locations (1):
- Kanazawa University, College of Medical Pharmaceutical and Health Sciences, School of Medicine, Department of Hematology, Kanazawa, Ishikawa-ken, Japan